CLINICAL TRIAL: NCT01786603
Title: Phase 2 Study of Rasagiline for Treatment of Amyotrophic Lateral Sclerosis
Brief Title: Rasagiline in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Richard Barohn, MD (Other)
Responsible Party: Sponsor-Investigator, Richard Barohn, MD, Gertrude and Dewey Zeigler Professor of Neurology and Chair, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12312; R01FD003739 (FDA)
Record Dates: First submitted 2012-11-28; First posted 2013-02-08 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rasagiline (Experimental): Rasagiline 1mg administered orally as a 2mg single dose once daily for 12 months.
  Interventions: Drug: Rasagiline
- Placebo (Placebo Comparator): Inactive ingredient equal to 1mg rasagiline 2mg administered as a single dose once daily for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rasagiline — Rasagiline 2mg once a day for 12 months.
  Other Names: Azilect
  Arms: Rasagiline
Drug: Placebo — Placebo (looks like study drug but has no active ingredients) once a day for 12 months.
  Arms: Placebo

SUMMARY:
ALS is a disorder that weakens motor strength and lung function. Rapid loss of motor neurons in the brain and spinal cord of ALS patients causes the symptoms of increasing weakness and loss of muscle function. Motor neurons are responsible for sending signals to muscles in our bodies to trigger movement. While there are drugs to help relieve symptoms of ALS, there is no cure for ALS.

Rasagiline is a drug with possible neuroprotective characteristics. Neuroprotective means that the nervous system may be protected against weakening. It is known that rasagiline has possible neuroprotective characteristics, but the effectiveness of rasagiline for patients with ALS has not been tested. Rasagiline is approved for the treatment of Parkinson's disease.

Rasagiline for treatment of ALS is not approved by the U.S. Food and Drug Administration (FDA) and is investigational. Investigational drugs are studied to find out if they are safe and effective in the treatment of diseases or conditions.

By doing this study, researchers hope to learn if rasagiline is safe and slows disease progression in patients with ALS.

Funding Source - FDA OOPD (FDA Orphan Products Division).

DETAILED DESCRIPTION:
The study is a phase II, double-blind, placebo-controlled, multicenter study of rasagiline 2mg/day. Subjects will be assigned to either active agent or placebo (3:1) for twelve months. Subjects will undergo outpatient evaluations at screening, baseline, and months 1, 2, 4, 6, 8, 10 and 12 and telephone assessments at months 3, 5, 7 and 9. There will be a close-out phone call 30 days post month 12.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of laboratory-supported probable, probable, or definite ALS, according to a modified El Escorial criteria, by the study investigator (Appendix IV).
2. 21 to 80 years of age inclusive.
3. VC greater or equal to 75% of predicted at screening and baseline.
4. Onset of weakness within 2 years prior to enrollment.
5. If patients are taking riluzole for ALS, they must be on a stable dose for at least thirty days prior to the baseline visit.
6. Women of childbearing age must be non-lactating and surgically sterile or using an effective method of birth control and have a negative pregnancy test.
7. Willing and able to give signed informed consent that has been approved by the Institutional Review Board (IRB).

Exclusion criteria

1. Requirement for tracheotomy ventilation or non-invasive ventilation for > 23 hours per day.
2. Patients on sympathomimetic agents. This includes pseudoephedrine, phenylephrine, phenylpropanolamine, and ephedrine.
3. Patients on analgesics with serotoninergic properties such as meperidine, tramadol, methadone and propoxyphene, flexeril.
4. Patients on fluoxetine or fluvoxamine.
5. Patients taking amitriptyline > 50 mg/d, trazodone and sertraline > 100 mg/d, citalopram > 20 mg/d or paroxetine > 30 mg/d.
6. Diagnosis of other neurodegenerative diseases (Parkinson disease, Alzheimer disease, etc).
7. Clinically significant history of unstable medical illness (unstable angina, advanced cancer, etc) over the last 30 days.
8. Has a diaphragm pacing device or plan on obtaining a diaphragm pacing device during the course of the study.
9. History of renal disease.
10. History of liver disease.
11. Current pregnancy or lactation.
12. Limited mental capacity such that the patient cannot provide written informed consent or comply with evaluation procedures.
13. History of recent alcohol or drug abuse or noncompliance with treatment or other experimental protocols.
14. Vital Capacity (VC) < 75% of predicted.
15. Receipt of any investigational drug within the past 30 days.
16. Women with the potential to become pregnant who are not practicing effective birth control.
17. Poorly controlled hypertensive subjects or resting systolic blood pressure (SBP) > 160 mmHg and/or diastolic (DBP) > 95 mmHg.
18. Use of BiPAP at screening.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-11-21 (Actual); Primary Completion 2016-07-27 (Actual); Study Completion 2016-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Barohn, MD, Principal Investigator — University of Kansas Medical Center
Locations (10):
- United States (10):
  - Phoenix Neurological Associates, Phoenix, Arizona
  - University of California - Irvine, Irvine, California
  - California Pacific Medical Center, San Francisco, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - St. Louis University, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Columbia University, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rasagiline | Placebo
Started | 60 | 20
Completed | 42 | 8
Not Completed | 18 | 12
Not completed — Death | 5 | 1
Not completed — Adverse Event | 6 | 2
Not completed — Physician decision to withdraw | 6 | 7
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rasagiline | Placebo | Total
Number analyzed (Participants) | 60 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (10.2) | 57.5 (8.5) | 57.95 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 7 | 27
  Male | 40 | 13 | 53

OUTCOME MEASURES:

1. Primary Outcome: ALS Functional Rating Scale-Revised (ALSFRS-R)
Description: Difference in ALS Functional Rating Scale - Revised (ALSFRS-R) score. The ALSFRS-R is an ordinal rating scale that assesses 12 functional activities. Each activity is scored between 0-4, with a total score ranging from 48 (normal function) to 0 (no function).
Time Frame: ALS Functional Rating Scale-Revised (ALSFRS-R) Difference from Baseline to Month 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Rasagiline | Placebo
Number analyzed (Participants) | 60 | 20
score on a scale | -1.00 [-1.22 to -0.77] | -1.26 [-1.64 to -0.87]

2. Secondary Outcome: Change in Vital Capacity (VC)
Description: Determine if decline in vital capacity is slower in participants taking 2 mg rasagiline than controls.
Time Frame: Vital Capacity Change from Baseline to Month 12
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Rasagiline | Placebo
Number analyzed (Participants) | 60 | 20
Liters | -2.24 [-2.86 to -1.64] | -2.48 [-3.54 to -1.43]

3. Secondary Outcome: Change in Quality of Life
Description: Participants completed the single-item ALSQOL (ALS Quality of Life) which asks participants to rank their global quality of life, considering all parts of their lives - physical, emotional, social, spiritual and financial - in the last 7 days and rate on a scale of 0 (very bad) to 10 (excellent).
Time Frame: Quality of Life Change from Baseline to Month 12
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Rasagiline | Placebo
Number analyzed (Participants) | 60 | 20
Score on a scale | -0.09 [-0.13 to -0.06] | -0.12 [-0.18 to -0.05]

4. Secondary Outcome: Number of Participants With Adverse Events
Description: Determine if participants on rasagiline 2 mg had a different safety profile than patients not on rasagiline. Adverse event information to be collected from date of enrollment until end of study participation.
Time Frame: Adverse Events from Baseline to Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Rasagiline | Placebo
Number analyzed (Participants) | 60 | 20
Participants | 28 | 15

5. Secondary Outcome: Difference in Survival Status Between Study Groups
Description: Determine if there is a difference in survival between participants on rasagiline than patients not on rasagiline
Time Frame: Survival status at Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Rasagiline | Placebo
Number analyzed (Participants) | 60 | 20
Participants | 55 | 19

6. Secondary Outcome: Effect of Study Drug on Apoptosis Markers
Description: Effect of rasagiline on the apoptosis markers (Annexin V stain) in participants with ALS. Assessed at baseline, month 6, and month 12; change from baseline to month 12 reported. Extra time point was not a pre-specified Primary or Secondary Outcome Measure.
Time Frame: Apoptosis Marker change from Baseline to Month 12
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Rasagiline | Placebo
Number analyzed (Participants) | 60 | 20
percentage of change | 0.019 (0.023) | 0.02 (0.019)

7. Secondary Outcome: Effect of Study Drug on Oxidative Stress
Description: Determine if oxygen radical antioxidant capacity is targeted by rasagiline in participants with ALS. Assessed at baseline, month 6, and month 12; change from baseline to month 12 reported. Extra time point was not a pre-specified Primary or Secondary Outcome Measure.
Time Frame: Oxidative Stress change from Baseline to Month 12
Measure: Mean (Standard Deviation); unit: pmole/ml
Arm/Group | Rasagiline | Placebo
Number analyzed (Participants) | 60 | 20
pmole/ml | 0.14 (0.73) | 1.21 (2.34)

ADVERSE EVENTS:
Arm/Group | Rasagiline | Placebo
All-Cause Mortality (participants affected / at risk) | 5/60 | 1/20
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/20
Other Adverse Events (participants affected / at risk) | 28/60 | 15/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rasagiline (N=60) | Placebo (N=20)
Cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Ear and Labyrinth (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eye (Eye disorders) | 3 (5) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 22 (49) | 12 (21)
General Disorders (General disorders) | 12 (20) | 3 (3)
Infections (Infections and infestations) | 11 (15) | 3 (4)
Injury, Poisoning, Procedural Complications (Injury, poisoning and procedural complications) | 11 (25) | 3 (4)
Laboratory Abnormality (Blood and lymphatic system disorders) | 6 (6) | 1 (1)
Metabolism and Nutrition (Metabolism and nutrition disorders) | 10 (11) | 3 (3)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 15 (25) | 9 (20)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Nervous System (Nervous system disorders) | 16 (20) | 6 (9)
Psychiatric (Psychiatric disorders) | 11 (19) | 6 (11)
Renal and Urinary (Renal and urinary disorders) | 8 (8) | 3 (3)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 15 (25) | 7 (10)
Skin (Skin and subcutaneous tissue disorders) | 5 (6) | 5 (7)
Surgical/Medical (Surgical and medical procedures) | 2 (2) | 2 (2)
Vascular (Vascular disorders) | 7 (10) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No